CLINICAL TRIAL: NCT01274871
Title: Late Sensory Changes From Chest Drain Insertion During Thoracotomy
Brief Title: Sensory Changes From Chest Drains
Status: Completed | Type: Observational
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: MD, Kim Wildgaard, Section for Surgical Pathophysiology 4074
Other Study IDs: H-B-2008-059/drain
Record Dates: First submitted 2011-01-11; First posted 2011-01-12 (Estimated); Last update posted 2011-01-12 (Estimated); Status verified 2011-01

CONDITIONS: Thoracotomy; Chronic Pain
Keywords: Thoracotomy; Chronic Pain; persistent post-surgical pain
MeSH Terms: conditions — Chronic Pain

STUDY DESIGN:
Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- lung cancer surgery

SUMMARY:
Does chest drains contribute to the post thoracotomy pain syndrome

ELIGIBILITY:
Inclusion Criteria:

* Age > 18
* Able to cooperate
* able to speak and read Danish

Exclusion Criteria:

* repeat surgery
* cognitive dysfunction
* other nerve injury on the thorax
* abuse (medicine/ alcohol etc)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Post thoracotomy patients after lung cancer in Denmark
Sampling Method: Non-Probability Sample
Enrollment: 21 (Actual)
Dates: Start 2009-12; Primary Completion 2010-04 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Pain (NRS) | 3 years postoperatively
Sensory thresholds | 3 years postoperatively

SECONDARY OUTCOMES:
Psychometrics (HADS) | 3 years

CONTACTS AND LOCATIONS:
Locations (1):
- Section for Surgical Pathophysiology 4074, Copenhagen, Denmark